CLINICAL TRIAL: NCT03380169
Title: Effectiveness in Preventing Surgical Site Infection by Using Prophylactic Occlusive Ionic Silver-containing Dressing in Abdominal Colorectal Surgery Patients - Randomized Controlled Trial
Brief Title: Preventing Surgical Site Infection by Using Prophylactic Occlusive Ionic Silver-containing Dressing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Princess Margaret Hospital, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Cheung Chi Yeung, Registered Nurse, Princess Margaret Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 61780111
Record Dates: First submitted 2017-11-02; First posted 2017-12-21 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: This is a single-blind two-arm parallel randomized controlled trial on occlusive ionic silver-containing dressing conducted in Princess Margaret Hospital (PMH). PMH is a major acute general hospital in Kowloon West Cluster in Hong Kong, providing 1,542 beds to maintain a wide range of specialist care. There are around 150 abdominal colorectal surgery provided every year in our department. Both the subjects, data collectors and outcome assessors will be blinded to the type of dressing being used. Eligible inpatients receiving colorectal surgery from the department of surgery will be consecutively recruited in each surgical ward (namely, A4 ward, B4 ward and CD4 ward).
Who Masked: Participant
Masking Description: Patients do not know which group they belongs to, and all wounds (for both experimental and control group) will be covered by gauze dressing at the top.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advance dressing (Experimental): Prophylactic advance wound dressing
  Interventions: Other: Prophylactic advance wound dressing
- Conventional gauze dressing (Active Comparator): Prophylactic conventional wound dressing
  Interventions: Other: Prophylactic conventional wound dressing

INTERVENTIONS:
Other: Prophylactic advance wound dressing — A combination of dressing including occlusive moist wound dressing to provide a barrier from the external environment and silver-containing dressing to reduce the inflammation of wounds and promotes healing
  Arms: Advance dressing
Other: Prophylactic conventional wound dressing — Conventional gauze dressing
  Arms: Conventional gauze dressing

SUMMARY:
Background: Ionic silver-containing dressing has been proven as a broad spectrum antimicrobial agent to reduce inflammation of wounds and promote healing. However, surgical incisions are usually dressed with conventional gauze dressing in colorectal surgery.

Objective: To compare the effectiveness in preventing surgical site infection (SSI) by using conventional gauze dressing and occlusive ionic silver-containing dressing.

Methods: This is a single-blind two-arm parallel randomized controlled trial on occlusive ionic silver-containing dressing conducted in Surgery Department of Princess Margaret Hospital. Two hundred patients who undergo emergency or elective abdominal colorectal surgery will be recruited and randomly assigned to have the surgical incisional wound dressed with conventional gauze dressing or occlusive ionic silver-containing dressing. Subjects will be assessed for SSI on day 3, 15 and 30 after operation in a clinical visit followed by phone interviews.

DETAILED DESCRIPTION:
Background Surgical site infections According to a Clean Care is safer programme by World Health Organization(WHO), the second most frequent and surveyed health care-associated infections in high-income countries is surgical site infections (SSI). The highest SSI is the colorectal surgery with 9.5% interlude per operations. SSI develop negative influence on patient outcome, such as burden the morbidity, mortality and extra expenses to health care system. The length of stay increased 9.7 days due to SSI in 2005 in USA, and more expenses spend on the antibiotics and the advanced dressing materials. Patient suffered from SSI will double the mortality rate in USA with increased cost and readmission for the treatment.

Modern dressing There are many different treatment and dressing options for health care providers for wound care. The dressings with advanced technology become more popular in recent days. Many studies show the importance of moist wound dressing to enhance the wound healing process. It can provide a moist wound environment, absorb the excess exudate, move away the microorganism and prevent their replication, and provide a barrier from the external environment than the conventional gauze dressing. Besides, a recommendation from the UK's National Institution for Health and Clinical Excellence (NICE) suggest that all surgical incision wound should be dressed with low-adhesive dressing for at least 3-5 days after operation. And a journal published in CINAHL Information System stated that the use of dressing with moist wound healing effects can help to reduce the SSI rate by 50% that the conventional gauze. On the other hand, there are studies commended that there are no significant different in prevention of SSI with the use of moist wound dressing. Therefore, it is a controversial issue on the effectiveness of preventing SSI by using moist wound dressing versus conventional gauze dressing.

Ionic silver-containing dressing Ionic silver (Ag+), is an active state silver oxidized biologically, is proved as a broad spectrum antimicrobial agent that is effective against aerobic, anaerobic, Gram-negative and Gram-positive bacteria, as well as fungi, viruses, and yeast with minimal development of bacterial resistance. Silver is used commonly in many dressings for the antimicrobial effect. Silver containing dressing can reduce the inflammation of wounds and promotes healing, since silver cations in the dressing can destroy microorganism by inactivating bacterial enzymes, disrupting the functions of cell membrane and binding the bacterial DNA/RNA to cause cell death and inhibiting cell replication.

Abdominal Colorectal surgery and ionic silver-containing dressing in Hong Kong In Hong Kong, colorectal cancer is the commonest cancer, there were around 5000 new cases in 2014. And it is the second leading cause of cancer deaths, in 2015, around colorectal cancer caused 2000 deaths. An unpublished internal audit carried out in surgical department in Princess Margaret Hospital (PMH) in 2015 found that the day 30 post-operation SSI incidence among patients with colorectal surgery using occlusive ionic silver-containing dressing (20%; 19/95) was statistically lower than those using conventional gauze dressing (52.9%; 9/17) with p=0.012 (Table 1). Although the effect of using silver dressing to reduce SSI rate is controversial, there are no formal study has been published locally. Therefore, it is meaningful to carry out a randomized controlled trial (RCT) to prove the significance of silver dressing in reduce SSI rate.

Objective To compare the SSI incidence among patients with abdominal colorectal surgery patients using prophylactic occlusive ionic silver-containing dressing and conventional gauze dressing.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or above undergo abdominal colorectal operation

Exclusion Criteria:

* Patients with cognitive impairment
* Patient with known allergic reactions to silver, hydrofibre or hydrocolloid
* Patient with non-closed wound immediate after operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-10-15 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
To assess if there are any surgical site infection on post-op day 30. | Post-op day 30
  Patient's case doctor will be responsible to document in date collection form, if there are surgical site infection occur. A research team is responsible for the data collection. The definition of surgical site infection will be according to CDC definitions of nosocomial surgical site infections: a modification of CDC definitions of surgical wound infection.

SECONDARY OUTCOMES:
To assess if there are any surgical site infection on Post-op day 3 & 15. | Post-op day 3 & 15
  Patient's case doctor will be responsible to document in date collection form, if there are surgical site infection occur. A research team is responsible for the data collection. The definition of surgical site infection will be according to CDC definitions of nosocomial surgical site infections: a modification of CDC definitions of surgical wound infection.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Yeung Cheung, BSc, Principal Investigator — Hospital Authority
Locations (1):
- Princess Margaret Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Field FK, Kerstein MD. Overview of wound healing in a moist environment. Am J Surg. 1994 Jan;167(1A):2S-6S. doi: 10.1016/0002-9610(94)90002-7. PMID 8109679
- [Background] Chen WY, Rogers AA, Lydon MJ. Characterization of biologic properties of wound fluid collected during early stages of wound healing. J Invest Dermatol. 1992 Nov;99(5):559-64. doi: 10.1111/1523-1747.ep12667378. PMID 1431216

DOCUMENTS (2):
  • Study Protocol (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT03380169/Prot_000.pdf
  • Informed Consent Form (2017-09-04): https://cdn.clinicaltrials.gov/large-docs/69/NCT03380169/ICF_001.pdf